CLINICAL TRIAL: NCT03901482
Title: EMERGE: A Randomized, Double-Blind, Parallel Group, Placebo-Controlled, Multicenter Study to Evaluate the Efficacy, Safety, and Tolerability of Single Doses of STS101 (Dihydroergotamine Nasal Powder) in the Acute Treatment of Migraine
Brief Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate STS101 in the Acute Treatment of Migraine
Acronym: EMERGE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Satsuma Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STS101-002
Record Dates: First submitted 2019-04-02; First posted 2019-04-03 (Actual); Results first posted 2023-06-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Migraine; Migraine With Aura; Migraine Without Aura
Keywords: dihydroergotamine; dihydroergotamine mesylate; migraine
MeSH Terms: conditions — Migraine Disorders; Migraine with Aura; Migraine without Aura | interventions — Dihydroergotamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- STS101 Low Dose (Experimental): STS101 (dihydroergotamine nasal powder), low dose
  Interventions: Drug: Dihydroergotamine
- STS101 High Dose (Experimental): STS101 (dihydroergotamine nasal powder), high dose
  Interventions: Drug: Dihydroergotamine
- STS101 Placebo (Placebo Comparator): STS101 Placebo
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Dihydroergotamine — Dihydroergotamine is a semi-synthetic derivative of ergotamine tartrate.
  Other Names: Dihydroergotamine Mesylate
  Arms: STS101 High Dose; STS101 Low Dose
Drug: Placebos — Placebo for STS101
  Other Names: STS101 Placebo
  Arms: STS101 Placebo

SUMMARY:
Study STS101-002 is a randomized, double-blind, parallel group, placebo-controlled, multicenter study to evaluate the efficacy, safety, and tolerability of single doses of STS101 (dihydroergotamine nasal powder) in the acute treatment of migraine

DETAILED DESCRIPTION:
The EMERGE trial is a multi-center, single-dose, randomized, double-blind, placebo-controlled, parallel group study in subjects with acute migraine (ages 18 to 65 years).

ELIGIBILITY:
Key Inclusion Criteria:

* Males or females, 18-65 years of age at the time of Screening Visit
* Subject has at least 1-year history of migraines (with or without aura), according to the International Classification of Headache Disorder, 3rd Edition (ICHD3)

Exclusion Criteria:

* Pregnant or breast-feeding women
* Women of child-bearing potential not using or not willing to use highly effective contraception.
* Diagnosis of headache conditions other than migraine with or without aura, including diagnosis of basilar or hemiplegic migraines or cluster headache.
* History of coronary artery disease, coronary artery vasospasm (including Printz-metals' angina), clinically significant arrhythmia or, peripheral vascular disease, ischemic disease (e.g. Raynaud's syndrome, ischemic bowel syndrome, angina pectoris, myocardial infarction, or documented silent ischemia); percutaneous coronary intervention, or cardiac surgery.
* History of cerebrovascular disease, including but not limited to stroke, transient ischemic attack, cerebral hemorrhage, subarachnoid hemorrhage.
* Diagnosis of major depression with current symptoms, psychosis, alcohol abuse or dependence, drug abuse or dependence, major psychiatric conditions (e.g. schizophrenia, psychosis or Bipolar disorder), dementia. Other significant neurological or psychiatric disorders (including other pain syndromes or risk of suicide) that in the opinion of the investigator might interfere with study participation and assessments or subject safety.
* Any clinically significant symptoms or conditions, including but not limited to central nervous system (e.g., seizures), cardiac, pulmonary, metabolic, renal, hepatic or gastrointestinal conditions or history of such conditions that, in the opinion of the investigator might interfere with study assessments or safety of participant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1201 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Detlef Albrecht, MD, Study Chair — Satsuma Pharmaceuticals, Inc.
Locations (117):
- United States (117):
  - Accel Clinical - Birmingham, Birmingham, Alabama
  - Alabama Clinical Therapeutics, Birmingham, Alabama
  - Alea Research, Phoenix, Arizona
  - Elite Clinical Studies, Phoenix, Arizona
  - Arizona Research Center, Phoenix, Arizona
  - Tucson Neuroscience Research, Tucson, Arizona
  - The Research Center of Southern California, Carlsbad, California
  - Med Center Medical Clinic, Carmichael, California
  - WR-PRI, Encino, California
  - Marvel Clinical Research, Huntington Beach, California
  - eStudySite, La Mesa, California
  - Collaborative Neuroscience, Long Beach, California
  - WP-PRI, Los Alamitos, California
  - Downtown LA Research, Los Angeles, California
  - Cal Neuro Research Group, Los Angeles, California
  - WR-PRI, Newport Beach, California
  - Alliance Sites, Oakland, California
  - Stanford Neuroscience Health Center, Palo Alto, California
  - National Research Institute, Panorama City, California
  - Empire Clinical Reserch, Pomona, California
  - Artemis Institute for Clinical Research- Riverside, Riverside, California
  - Artemis Institute of Clinical Research - San Diego, San Diego, California
  - Pacific Research Network, San Diego, California
  - WR-MCCR, San Diego, California
  - Optimus Medical Group, San Francisco, California
  - Artemis Institute for Clinical Research- San Marcos, San Marcos, California
  - Neurological Research Institute, Santa Monica, California
  - Schuster Medical Research Institute, Sherman Oaks, California
  - Southern California Research, Simi Valley, California
  - Encompass Clinical Research, Spring Valley, California
  - Hartford Headache Center, East Hartford, Connecticut
  - CMR of Greater New Haven, Hamden, Connecticut
  - New England Institute for Neurology and Headache, Stamford, Connecticut
  - Chase Medical Research, Waterbury, Connecticut
  - Accel Clinical - DeLand, DeLand, Florida
  - Gulf Coast Clinical Research, Fort Myers, Florida
  - MD Clinical, Hallandale, Florida
  - AGA Clinical Trials, Hialeah, Florida
  - Galiz Research- Hialeah, Hialeah, Florida
  - Research Centers of America, Hollywood, Florida
  - CNS Healthcare, Jacksonville, Florida
  - Multispecialty Research Associates, Lake City, Florida
  - ClinCloud, Maitland, Florida
  - Premier Clinical Reserch Institute, INC, Miami, Florida
  - QPS MRA, Miami, Florida
  - Applemed Research Group, Miami, Florida
  - Biotech Pharmaceuticals Group, Miami, Florida
  - Behavioral Clinical Research, North Miami, Florida
  - Sensible Health, Ocoee, Florida
  - Accel - Orange City, Orange City, Florida
  - CNS Health Care - Orlando, Orlando, Florida
  - Neurology Associates of Ormond Beach, Ormond Beach, Florida
  - Infinity Clinical Research, LLC, Sunrise, Florida
  - Precision Clinical Research, Sunrise, Florida
  - Clinical Research CF, Winter Haven, Florida
  - Conquest Research, Winter Park, Florida
  - Neuro Studios, Decatur, Georgia
  - Advanced Clinical Research, Meridian, Idaho
  - PMG Research of DuPage Medical Group, Downers Grove, Illinois
  - Healthcare Research Network II, LLC, Flossmoor, Illinois
  - Phoenix Medical Reserch, Prairie Village, Kansas
  - Delricht - Baton Rouge, Baton Rouge, Louisiana
  - Tandem Clinical Research, Marrero, Louisiana
  - Delricht - NewOrleans, New Orleans, Louisiana
  - Boston Clinical Trials, Boston, Massachusetts
  - BTC of New Bedford, New Bedford, Massachusetts
  - Medvadis Research Group, Watertown, Massachusetts
  - Michigan Headache and Neurological Institute, Ann Arbor, Michigan
  - Michigan Pain Consultants, Wyoming, Michigan
  - Minneapolis Clinic of Neurology, Burnsville, Minnesota
  - StudyMetrix Research, City of Saint Peters, Missouri
  - Healthcare Research Network II, LLC, Hazelwood, Missouri
  - Clinvest Research, Springfield, Missouri
  - Montana Medical Research, Missoula, Montana
  - Quality Clinical Research, Omaha, Nebraska
  - Altea Research, Las Vegas, Nevada
  - Wake Research-Clinical Research Center of Nevada, Las Vegas, Nevada
  - Clinical Research of South Nevada, Las Vegas, Nevada
  - Dartmouth-Hitchcock Clinical Trials Office, Lebanon, New Hampshire
  - Hassman Research Institute, Berlin, New Jersey
  - Albuquerque Clinical Trials, Albuquerque, New Mexico
  - Albuquerque Neuroscience, Albuquerque, New Mexico
  - SPRI Clinical Trials, Brooklyn, New York
  - Manhattan Behavioral Medicine, New York, New York
  - Rochester Clinical Research, Rochester, New York
  - Montefiori Medical Center, The Bronx, New York
  - Upstate Clinical Research Associates, Williamsville, New York
  - Headache Wellness Center - Greensboro, Greensboro, North Carolina
  - PharmQuest, Greensboro, North Carolina
  - M3-Wake Research, Raleigh, North Carolina
  - PMG Research of Wilmington, Wilmington, North Carolina
  - Lillestol Research, Fargo, North Dakota
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Rapid Medical Research Inc., Cleveland, Ohio
  - Aventiv Research, Columbus, Ohio
  - Neurology Diagnosis, Dayton, Ohio
  - Delynn Institute, Oklahoma City, Oklahoma
  - Delricht Research, Tulsa, Oklahoma
  - Thomas Jefferson University/Jefferson Headache Center, Philadelphia, Pennsylvania
  - CNS Research Inc - Rhode Island, Rumford, Rhode Island
  - Omega Medical Research, Warwick, Rhode Island
  - WR-ClinSearch, Chattanooga, Tennessee
  - CNS Healthcare, Memphis, Tennessee
  - Clinical Research Associates, Nashville, Tennessee
  - Nashville Neuroscience Group, Nashville, Tennessee
  - Wellness Clinical Research, Allen, Texas
  - FutureSearch Trials of Neurology, Austin, Texas
  - Future Search Trials, Dallas, Texas
  - HRMD Research, Dallas, Texas
  - Texas Center for Drug Development, Houston, Texas
  - SMS Clinical Research, Mesquite, Texas
  - DM Clinical Research, Tomball, Texas
  - ClinPoint Trials, Waxahachie, Texas
  - Aspen Clinical Research, Orem, Utah
  - Wasatch Clinical Research, Salt Lake City, Utah
  - Highland Clinical Research, Salt Lake City, Utah
  - Charlottesville Medical Research, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 119 sites in the United States.
Pre-assignment Details: A total of 1201 participants were randomized in the study, of which 1065 reported a qualifying migraine attack, received study drug, and reported a post-dose efficacy evaluation for at least one time point at or before the 2-hour timepoint (mITT population).
Groups:
- STS101 Low Dose: Subjects received a single oral dose of STS101 (dihydroergotamine nasal powder) 3.9 mg.
- STS101 High Dose: Subjects received a single oral dose of STS101 (dihydroergotamine nasal powder) 5.2 mg.
- STS101 Placebo: Subjects received a single oral dose of Placebo for STS101 (dihydroergotamine nasal powder).
Period: Overall Study
Arm/Group | STS101 Low Dose | STS101 High Dose | STS101 Placebo
Started | 399 | 400 | 402
Completed | 363 | 368 | 364
Not Completed | 36 | 32 | 38

BASELINE CHARACTERISTICS:
Population: Patient demographics are presented for the safety population defined as all subjects who were randomized and received the study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | STS101 Low Dose | STS101 High Dose | STS101 Placebo | Total
Number analyzed (Participants) | 363 | 367 | 363 | 1093
Age, Customized [Count of Participants; unit: Participants]
  Age Group (n (%)): 18-35 years | 123 | 117 | 122 | 362
  Age Group (n (%)): >30-50 years | 164 | 186 | 176 | 526
  Age Group (n (%)): >50-65 years | 76 | 64 | 65 | 205
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 318 | 320 | 317 | 955
  Male | 45 | 47 | 46 | 138
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 3 | 7
  Asian | 6 | 12 | 13 | 31
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 1 | 4
  Black or African American | 55 | 60 | 41 | 156
  White | 293 | 292 | 304 | 889
  More than one race | NA — No data was collected for more than one race. | NA — No data was collected for more than one race. | NA — No data was collected for more than one race. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported | 4 | 1 | 1 | 6
Region of Enrollment [Number; unit: participants]
  United States | 363 | 367 | 363 | 1093

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Freedom From Migraine Headache Pain at 2 Hours Post Dose
Description: The subject's rating was documented on a four-point scale from no pain (= 0), mild pain (= 1), moderate pain (= 2) to severe pain (= 3). Pain freedom means the pain went from moderate (2) or severe (3) to no pain (0).
Time Frame: 2 Hours Post-Dose
Population: The analysis was performed on the mITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | STS101 Low Dose | STS101 High Dose | STS101 Placebo
Number analyzed (Participants) | 354 | 353 | 358
Participants | 69 | 68 | 53

2. Primary Outcome: Percentage of Subjects With Freedom From Most-Bothersome Symptom at 2 Hours Post Dose
Description: Subjects were prompted to document the presence of 3 symptoms (photophobia, phonophobia, and nausea) immediately before study drug administration and during the treated migraine attack.
Time Frame: 2 Hours Post-Dose
Population: This analysis was conducted on the mITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | STS101 Low Dose | STS101 High Dose | STS101 Placebo
Number analyzed (Participants) | 354 | 353 | 358
Participants | 133 | 139 | 119

3. Secondary Outcome: Percentage of Subjects With Relief From Migraine Headache Pain at 2 Hours Post Dose
Description: The subject's rating was documented on a four-point scale from no pain (= 0), mild pain (= 1), moderate pain (= 2) to severe pain (= 3). Pain relief means the pain went from moderate (2) or severe (3) to mild pain (1) or no pain (0).
Time Frame: 2 Hours Post Dose
Population: This analysis was conducted on the mITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | STS101 Low Dose | STS101 High Dose | STS101 Placebo
Number analyzed (Participants) | 354 | 353 | 358
Participants | 180 | 177 | 166

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) were collected from informed consent up to the end of study, and adverse events (AEs) were collected from randomization up to the end of the study (7±3 days after migraine treatment or early study termination).
Description: The safety population was used for adverse event reporting.
Arm/Group | STS101 Low Dose | STS101 High Dose | STS101 Placebo
All-Cause Mortality (participants affected / at risk) | 0/363 | 0/367 | 0/363
Serious Adverse Events (participants affected / at risk) | 0/363 | 1/367 | 0/363
Other Adverse Events (participants affected / at risk) | 49/363 | 52/367 | 19/363
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | STS101 Low Dose (N=363) | STS101 High Dose (N=367) | STS101 Placebo (N=363)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — The subject was hospitalized for pneumonia after study randomization but before use of study medication.
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | STS101 Low Dose (N=363) | STS101 High Dose (N=367) | STS101 Placebo (N=363)
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 20 (20) | 21 (21) | 7 (7)
Dyseusia (Nervous system disorders) | 15 (15) | 18 (18) | 5 (5)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 5 (5) | 4 (4)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 8 (8) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-09): https://cdn.clinicaltrials.gov/large-docs/82/NCT03901482/Prot_SAP_000.pdf